CLINICAL TRIAL: NCT01866839
Title: Peripheral Blood Stem Cell Allotransplantation For Hematological Malignancies Using Ex Vivo CD34 Selection - a Platform For Adoptive Cellular Therapies
Brief Title: Preventing Stem Cell Transplant Complications With a Blood Separator Machine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130144; 13-H-0144
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2018-06-28

CONDITIONS: MDS (Myelodysplastic Syndrome); Myeloproliferative Disorder; Lymphoma, Non-Hodgkin; ALL (Acute B-Lymphoblastic Leukemia); AML (Acute Myelogenous Leukemia
Keywords: Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Chronic Lymphocytic Leukemia (CLL); Chronic Myelogenous Leukemia (CML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CD34+ cell positively selected graft stem cell recipient (Experimental): Recipients received a myeloablative conditioning regimen of cyclophosphamide (120 mg/kg total), fludarabine (125 mg/m2 total) and total body irradiation (1200 cGy with lung shielding to 600 cGy), followed by an infusion of a stem cell product selected for CD34+ progenitors using the Miltenyi CliniMACS® system. Older subjects will receive a lower dose of irradiation (800 or 600 cGy based on age) to reduce the regimen intensity.
  Interventions: Device: Graft Manipulation (CD34+ Selection)

INTERVENTIONS:
Device: Graft Manipulation (CD34+ Selection)

SUMMARY:
Background:

- Researchers are working to make stem cell transplant procedures safer and more effective. One complication of transplants is graft-versus-host disease (GVHD). This complication happens when certain white blood cells from the donor attack the recipient's own body. Researchers want to test a blood separator machine that may help remove more of the donor's white blood cells before transplant. They will study donors and recipients during stem cell transplant to see how well this process can prevent GVHD and other complications.

Objectives:

- To see if a new blood separator machine can improve outcomes of stem cell transplants.

Eligibility:

* Individuals between 10 and 75 years of age who are having a stem cell transplant for leukemia or other blood-related cancers.
* Donors for the stem cell transplant.

Design:

* Recipients and donors will be screened with a physical exam and medical history.
* Donors will have two blood collection procedures. The first will collect only white blood cells, and return the rest of the blood. After the first collection, participants will have filgrastim injections to help their stem cells enter their blood. Then, they will have a second blood collection for the stem cells.
* Recipients will have radiation and chemotherapy to prepare for the stem cell transplant. They will then have the stem cell transplant with the donor cells that have been treated with the blood separator machine.
* Recipients will be monitored closely after the procedure. They may receive some of their donor's white blood cells if needed to fight serious infections.
* Recipients will have the regular standard of care after their transplant. Blood samples will be taken and any side effects will be monitored and treated.

DETAILED DESCRIPTION:
Peripheral blood stem cell transplant research carried out by the NHLBI BMT Unit focus on transplant techniques designed to decrease graft versus host disease (GVHD), increase the graft-versus-leukemia (GVL) effect and reduce the risk of post-transplant graft rejection.

Through incremental transplant clinical trials we have shown that by controlling the stem cell (CD34+ cell) and T lymphocyte (CD3+ cell) dose, severe GVHD can be reduced whilst beneficial GVL effects can be preserved. We found that T cell depleted transplants using the Nexell/Baxter Isolex 300i system and subsequently, the Miltenyi CliniMACS[registered] CD34+ system to obtain high CD34+ doses depleted of lymphocytes were safe to administer and associated with less severe acute GVHD and promising response rates and overall survival. Our previous trials have helped us to create the transplant environment (significant lymphodepletion and minimal post transplant immunosuppression) that make for an ideal platform for adoptive cellular immunotherapy. Adoptive cell transfer is the passive transfer of immune cells, into a new recipient host with the goal of transferring the immunologic functionality and characteristics into the new host.

This protocol is designed to evaluate the safety and efficacy of the Miltenyi CliniMACS[registered] CD 34 selection system in HLA-matched sibling allogeneic peripheral blood stem cell transplant. The manipulation of the graft is the primary research intervention, subject to IDE# 15632, and all other aspects of clinical management on this protocol are standard care. The target CD34+ dose range will be >3 x 10(6)/kg and the target CD3+ dose range will be 5 x 10(4)/kg to 1 x 10(6)/kg. Once we demonstrate adequacy of this platform for engraftment and absence of significant GVHD in ten consecutive recipients, we will seek IRB permission to proceed with planned adoptive cellular therapies.

The protocol will accrue up to 96 transplant recipients aged 10-80 with a hematological malignancy and their HLA-matched sibling donors, in whom allogeneic stem cell transplantation from an HLA-matched sibling would be routinely indicated. Diagnostic categories will include acute and chronic leukemia, myelodysplastic syndromes, lymphomas, multiple myeloma and myeloproliferative syndromes.

Subjects will receive a myeloablative conditioning regimen of cyclophosphamide (120 mg/kg total), fludarabine (125 mg/m(2) total) and total body irradiation (1200 cGy with lung shielding to 600 cGy), followed by an infusion of a stem cell product selected for CD34+ progenitors using the Miltenyi CliniMACS[registered] system. Older subjects will receive a lower dose of irradiation (800 or 600 cGy based on age) to reduce the regimen intensity.

The overall objective is to assess the feasibility of using this system as a platform for cellular immunotherapy initiatives. The primary study endpoint will be overall survival at day +200. Stopping criteria for safety will monitor non-relapse mortality at day +200 and late disease free survival at 2 years. Secondary endpoints will be standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD and relapse of disease.

ELIGIBILITY:
* INCLUSION CRITERIA RECIPIENT

5.1.1 Ages 10-80 years inclusive

5.1.2 Any one of the following hematologic conditions, confirmed by pathology, meeting a standard indication for allogeneic stem cell transplant:

5.1.2.1 Chronic myelogenous leukemia (CML): Subjects under the age of 21 in chronic phase OR Subjects ages 10-80 in chronic phase who have failed or are intolerant to treatment with second generation tyrosine inhibitors OR Subjects ages 10-80 in accelerated phase or blast transformation. OR

5.1.2.2 Acute lymphoblastic leukemia (ALL): any of these categories: Adult ALL including standard risk; Pediatric ALL in first remission with high-risk features (presenting leukocyte count >100,000/cu mm, karyotypes t(9; 22), t4, t19, t11, biphenotypic leukemia). All second or subsequent remissions, primary induction failure, partially responding or untreated relapse. OR

5.1.2.3 Acute myelogenous leukemia (AML): AML in first remission - except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), c-kit unmutated AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse. OR

5.1.2.4 Myelodysplastic syndromes(MDS): any of these categories - refractory anemia with transfusion dependence, refractory anemia with ANC<500/microL, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia, atypical MDS/myeloproliferative syndromes. OR

5.1.2.5 Myeloproliferative disorders including atypical (Ph-negative) chronic myeloid and neutrophilic leukemias, progressing myelofibrosis, and polycythemia vera, essential thrombocythemia either in transformation to acute leukemia or with progressive transfusion requirements or pancytopenia. OR

5.1.2.6 Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000 / microl) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy. OR

5.1.2.7 Non-Hodgkin s lymphoma including Mantle cell lymphoma relapsing or refractory to standard of care treatments. OR

5.1.2.8 Multiple myeloma, Waldenstroms macroglobulinemia, unresponsive or relapsed following standard of care treatments. OR

5.1.2.9 Hodgkin's Lymphoma relapsing following an autologous transplant. OR

5.1.2.10 Other rare hematologic malignancies for which hematopoietic stem cell transplantation has been performed and offers a durable remission or as the only option for potential for cure.

* Chemotherapy-resistant multisystem Langerhans cell histiocytosis (MSLCH) especially involving organs like the bone marrow, liver, spleen, and lungs
* Aggressive systemic mastocytosis, and mast cell leukemia (MCL) in first CR (CR1)
* Hypereosinophilic syndrome who have failed imatinib therapy or FIP1L1-PDGFRa-negative patients who develop end-organ dysfunction
* Adult T-cell leukemia/lymphoma at first diagnosis
* Refractory or disseminated nasal-type extranodal NK/T-lymphoma or aggressive Natural killer cell leukemia/lymphoma
* Mycosis fungoides and S(SqrRoot)(Copyright)zary syndrome after failure of two or three initial therapies
* Primary or relapsed refractory Angioimmunoblastic T-cell lymphoma at first diagnosis
* Hepatosplenic T-cell lymphoma (gamma/delta T-cell lymphoma) at first diagnosis
* T-cell prolymphocytic leukemia at first diagnosis
* Subcutaneous panniculitic T-cell lymphoma at first diagnosis
* Hematodermic neoplasm (blastic natural killer cell lymphoma or Blastic plasmacytoid dendritic cell neoplasm) at first diagnosis

5.1.3 HLA identical (6/6) related donor.

5.1.4 For adults: ability to comprehend the investigational nature of the study and provide informed consent. For minors: written informed consent from one parent or guardian. Informed oral assent from minors: the process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA RECIPIENT (any of the following)

5.2.1 Major anticipated illness or organ failure incompatible with survival from transplant

5.2.2 Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and making informed consent impossible.

5.2.3 Positive pregnancy test for women of childbearing age

5.2.4 DLCO adjusted for Hb and ventilation< 50% predicted

5.2.5 Left ventricular ejection fraction < 40% (evaluated by ECHO) or < 30% (evaluated by MUGA)

5.2.6 AST/SGOT > 10 times ULN

5.2.7 Total bilirubin > 5 times ULN

5.2.8 Estimated GFR < 15 mL/min

5.2.9 Recipients who have active infections with HIV or active hepatitis C (HCV)

INCLUSION CRITERIA DONOR

5.3.1 Related donor, HLA identical (6/6) with recipient

5.3.2 Weight greater than or equal to 18 kg

5.3.3 Age greater than or equal to 2 or less than or equal to 80 years old

5.3.4 For adults: ability to comprehend the investigational nature of the study and provide informed consent. For minors: written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA DONOR (any of the following)

5.4.1 Pregnant or breast-feeding. Lactating donors are permitted provided breast milk is discarded during the days filgrastim (G-CSF) is given

5.4.2 Unfit to receive G-CSF and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension)

5.4.3 Sickling hemoglobinopathy including HbSS, HbSC

5.4.4 Donors who are positive for HIV, active hepatitis B (HBV), hepatitis C (HCV) or human Tcell lymphotropic virus (HTLV-I/II)

5.4.5 Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the donation process unlikely, and making informed consent impossible.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-05-29; Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sawa Ito, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armitage JO. Bone marrow transplantation. N Engl J Med. 1994 Mar 24;330(12):827-38. doi: 10.1056/NEJM199403243301206. No abstract available. PMID 8114836
- [Background] Barrett AJ. Graft-versus-host disease: basic considerations. Recent Results Cancer Res. 1993;132:185-95. doi: 10.1007/978-3-642-84899-5_19. No abstract available. PMID 8265860
- [Background] Appelbaum FR. Haematopoietic cell transplantation as immunotherapy. Nature. 2001 May 17;411(6835):385-9. doi: 10.1038/35077251. PMID 11357147

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant signed consent but did not start study
Period: Overall Study
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Started | 40
Completed | 30
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 32
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 4
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Secondary Outcome: Disease Free Survival at 2 Years
Description: Disease Free Survival at 2 years
Time Frame: 2 years
Population: Subjects for whom the Miltenyi CliniMACS CD34 selection system was used for graft manipulation in HLA-matched sibling allogeneic stem cell transplantation
Measure: Number; unit: percentage of participant
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
percentage of participant | 60.8

2. Secondary Outcome: Disease Progression
Description: Incidence of relapse / disease progression
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 11

3. Secondary Outcome: Incidence of Acute GVHD
Description: Participants who develop acute GVHD
Time Frame: 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 26

4. Secondary Outcome: Incidence of Chronic GVHD
Description: Participants who develop chronic GVHD
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 14

5. Secondary Outcome: Median Time to ANC>500/mm3
Description: Time in days
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Days | 12 [9 to 28]

6. Secondary Outcome: Median Time to Platelets>20K/mm3
Description: Time in days
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Days | 15 [14 to 28]

7. Primary Outcome: Overall Survival
Description: Determine the rate of overall survival at 200 day
Time Frame: 200 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 36

8. Secondary Outcome: Severity of Acute GVHD
Description: Grade I
Time Frame: 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 10

9. Secondary Outcome: Severity of Acute GVHD
Description: Grade II
Time Frame: 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 7

10. Secondary Outcome: Severity of Acute GVHD
Description: Grade III
Time Frame: 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 8

11. Secondary Outcome: Severity of Acute GVHD
Description: Grade IV
Time Frame: 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 1

12. Secondary Outcome: Severity of Chronic GVHD
Description: Extensive
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 10

13. Secondary Outcome: Severity of Chronic GVHD
Description: Limited
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
Number analyzed (Participants) | 40
Participants | 4

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | CD34+ Cell Positively Selected Graft Stem Cell Recipient
All-Cause Mortality (participants affected / at risk) | 11/40
Serious Adverse Events (participants affected / at risk) | 38/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD34+ Cell Positively Selected Graft Stem Cell Recipient (N=40)
Anaemia (Blood and lymphatic system disorders) | 1
Engraftment syndrome (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiomyopathy acute (Cardiac disorders) | 1
Diastolic dysfunction (Cardiac disorders) | 1
Fluid overload (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Clostridium difficile colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cytomegalovirus gastrointestinal infection (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastroenteritis astroviral (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Viral diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adult failure to thrive (General disorders) | 1
Catheter site pain (General disorders) | 1
Drug withdrawal convulsions (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Incarcerated hernia (General disorders) | 1
Pain (General disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 7
Acute graft versus host disease in skin (Immune system disorders) | 3
Chronic graft versus host disease (Immune system disorders) | 1
Chronic graft versus host disease in intestine (Immune system disorders) | 3
Food allergy (Immune system disorders) | 1
Reaction to preservatives (Immune system disorders) | 1
Transplant rejection (Immune system disorders) | 1
Adenovirus infection (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 6
BK virus infection (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 5
Cystitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 7
Epstein-Barr viraemia (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 3
Escherichia sepsis (Infections and infestations) | 2
Fungaemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia fungal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Salmonella sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 1
Stenotrophomonas infection (Infections and infestations) | 1
suspected infection (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Varicella zoster virus infection (Infections and infestations) | 1
Vulvovaginal human papilloma virus infection (Infections and infestations) | 1
Wound abscess (Infections and infestations) | 1
Delayed engraftment (Injury, poisoning and procedural complications) | 1
Engraft failure (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Procedural headache (Injury, poisoning and procedural complications) | 1
Anion gap (Investigations) | 1
Body temperature increased (Investigations) | 12
Hyperkalaemia (Investigations) | 1
Headache (Nervous system disorders) | 1
Orthostatic hypotension (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Altered state of consciousness (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis management (Surgical and medical procedures) | 1
Orthostatic hypotension (Vascular disorders) | 1
Syncope (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
1 participant signed consent but did not start study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT01866839/Prot_SAP_000.pdf